CLINICAL TRIAL: NCT06988384
Title: Effects of a Professional Objective Bike Fit on Power Output and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, River Falls (Other)
Responsible Party: Principal Investigator, Gregory Ruegsegger, Associate Professor, University of Wisconsin, River Falls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FY2024-7
Record Dates: First submitted 2025-05-07; First posted 2025-05-23 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy Population
Keywords: bike fitting; bike configuration; peak power; functional threshold power; cycling pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- idmatch bike fitting (Experimental): Participants will undergo bike fitting using the idmatch system, which utilizes three-dimensional motion capture to optimize rider position.
  Interventions: Other: Bike fitting

INTERVENTIONS:
Other: Bike fitting — Participants underwent bike fitting using the idmatch system, which utilizes three-dimensional motion capture to optimize rider position.

SUMMARY:
This study aims to evaluate whether an objective, data-driven bike fitting using the id match 3D motion capture system improves power output in recreational cyclists. Participants will complete two cycling performance tests, a 6-second Wingate Anaerobic Test (PPT6) and a 20-minute Functional Threshold Power (FTP) test, before and after receiving a professional bike fitting. The primary outcome is the change in power output on both tests. Secondary outcomes include subjective measures of comfort, pain, and perceived exertion. The goal is to determine whether bike fitting alone, independent of training, can enhance both performance and the overall riding experience.

DETAILED DESCRIPTION:
This is a prospective, interventional crossover study evaluating the impact of professional bike fitting on cycling performance and comfort in recreational cyclists. All participants must engage in structured physical activity at least twice per week (≥30 minutes per session), own a road or gravel bicycle, and are available for two laboratory visits within a 96-hour period. All participants must complete the PAR-Q+ and a health history questionnaire.

At Visit 1, participants will undergo baseline testing. Their current bike setup will be replicated on a Wattbike ergometer. Participants will complete two performance tests: a six-second peak power test (PPT6) and a 20-minute Functional Threshold Power (FTP) test. For the PPT6, participants perform a seated sprint from a dead stop following a five-minute warm-up and two-minute rest. Metrics collected include peak power (W), relative peak power (W/kg), cadence (rpm), and leg imbalance (%). The FTP test will be conducted on each participant's personal bicycle mounted to a Wahoo KICKR MOVE smart trainer. Power, cadence, and torque are recorded, along with physiological data captured using a Polar H10 heart rate monitor and a COSMED Quark CPET system to measure VO₂, VCO₂, and RER. Following these assessments, participants will receive a professional bike fitting using the id match Smart Bike system.

The id match system (Casella d'Asolo, Italy) uses 3D motion capture, static anthropometric scans (e.g., limb length, lumbar flexion, foot dimensions), and machine learning algorithms to optimize rider positioning. The fitting process adjusts variables such as saddle height, saddle setback, handlebar reach and drop, and cleat position. A certified id match fitter will perform each fitting, which is guided by participant-reported cycling history and pain ratings by body region on a 1-10 scale.

Between 48 and 96 hours after the initial visit, participants will return for Visit 2 and repeat both the PPT6 and FTP tests using their updated bike configuration. All equipment, testing protocols, and data collection methods remain consistent between visits.

Primary outcome measures include peak power and relative peak power (W/kg) from the PPT6, and FTP (W), relative FTP (W/kg), and average torque (ft-lb.) from the 20-minute FTP test. Secondary outcomes include perceived exertion (Borg RPE 6-20 scale), discomfort (Likert scale 1-20), region-specific pain, and biomechanical changes to bike setup (e.g., saddle height, setback, cleat position, joint angles).

ELIGIBILITY:
Inclusion Criteria:

Participates in structured exercise more than 2 times per week (≥ 30 minutes per session) Owns a road or gravel bicycle Available for two laboratory visits within a 96-hour period Passes the PAR-Q+ questionnaire

Exclusion Criteria:

Has previously undergone a professional bicycle fitting

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Power output | Baseline (Day 1) and 48 to 96 hours post-baseline
  Peak power during a six-second peak power test
Functional threshold power | Baseline (Day 1) and 48 to 96 hours post-baseline
  Aveage power during a 20-minute functional threshold power test.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Ruegsegger, Ph.D., Principal Investigator — University of Wisconsin, River Falls
Locations (1):
- University of Wisconsin - River Falls, River Falls, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data related to primary and secondary outcomes will be shared. This includes pre- and post-fitting results from the 6-second Wingate Anaerobic Test (peak power), the 20-minute Functional Threshold Power (average power and torque), and self-reported measures of perceived exertion and musculoskeletal discomfort. Basic demographic data (age, sex, height, weight, cycling experience) will also be included.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be made available within 6 months of publication of the primary results and will remain available for up to 3 years following publication.
Access Criteria: Data will be available to qualified researchers for non-commercial academic purposes. Requests must include a methodologically sound proposal and will be reviewed by the study investigators. Data requestors must agree to a data use agreement to ensure participant confidentiality.